CLINICAL TRIAL: NCT06413641
Title: VIsualization of Coronary Artery Disease for Modification of RISK Factors. Prevention of Disease Progression in Patients With Non-Obstructive Coronary Atherosclerosis.
Brief Title: VIsualization of Coronary Artery Disease for Modification of RISK Factors
Acronym: VICAD-RISK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other); Vejle Hospital (Other); Gødstrup Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Bjarne Linde Nørgaard, MD, Professor, DMSCi, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NNF21OC0068200; 1-10-72-213-22 (Other: VMK NVK)
Record Dates: First submitted 2024-04-12; First posted 2024-05-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Non-Obstructive Coronary Atherosclerosis
Keywords: Coronary computed tomography; Hypercholesterolemia
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1:1 to post-CTA usual care follow up in general practice or one of two intervention strategies ("low" or "high" intensity intervention). Patients randomized to the intervention groups will be invited to an individualized video-based or ambulatory consultation by a special trained nurse within 2 weeks from the index CTA test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Active Comparator): Usual care follow up in general practice
  Interventions: Other: Follow up at general practice
- Low intensity intervention (Experimental): Individualized video-based or ambulatory consultation by a special trained nurse within 2 weeks from the index CTA test
  Interventions: Other: Consultation
- High intensity intervention (Experimental): Individualized video-based or ambulatory consultation by a special trained nurse within 2 weeks from the index CTA test combined with visualization of the individual CTA images with focus on the atherosclerotic findings and the effect of statin treatment on the disease
  Interventions: Other: Consultation; Other: Visualization of CTA images

INTERVENTIONS:
Other: Follow up at general practice — As described before
  Arms: Usual care
Other: Consultation — As described before
  Arms: High intensity intervention; Low intensity intervention
Other: Visualization of CTA images — As described before
  Arms: High intensity intervention

SUMMARY:
The VICAD-RISK study assesses if visualization of coronary CT angiography (CTA) images in participants with non-obstructive coronary artery disease will improve LDL lowering, reduce reporting of side effects by cholesterol lowering medications, and modify the coronary artery disease phenotype over 12 months.

DETAILED DESCRIPTION:
In Denmark non-obstructive coronary artery disease is found in 35-40% of patients undergoing coronary CT angiography for suspected coronary artery disease. Modification of risk factors is essential in patients with coronary artery disease to prevent major cardiovascular events. However, in non-obstructive coronary artery disease, initiation and adherence to treatment with lipid lowering therapy is poor.

The study will include 273 patients from 5 different sites; patients will be randomized into 3 groups; standard follow up by general practice, structured disease education or the combination of the latter with visualization of coronary CT angiography images. A follow-up CT angiography will be performed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of nonobstructive coronary artery disease
* No known coronary artery disease (no previous coronary revascularization)
* CAD-Rads score 1-3
* LDL cholesterol > 2.0 mmol/l
* Life expectancy >3 years
* Signed informed consent

Exclusion Criteria:

* Post CTA test indication for invasive coronary angiography
* Non-evaluable CTA exam
* Obstructive coronary disease (One or more coronary stenosis ≥70%, left main >40%)
* Ongoing lipid lowering medical treatment (Patients already on lipid lowering medical therapy can be included if the treatment was initiated <3 months before the time of the CTA test)
* BMI >40
* Renal insufficiency (eGFR <40 ml/min)
* Allergy to iodinated contrast media
* Contraindications to statins (Active liver disease Child-Pugh A, B and C, excessive alcohol consumption)
* Participation in a cardiac rehabilitation or lifestyle modification program
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in LDL cholesterol | 12 months
  Assessed by measurement of LDL cholesterol level (mmol/L) in blood samples at baseline and 12 months follow-up

SECONDARY OUTCOMES:
Side effects of statin therapy | 12 months
  Assessed with questionnaire (based on numeric pain rating scale) at 3 and 12 months follow-up
Changes in high risk coronary plaque volumes | 12 months
  Assessed by changes in the CT-derived coronary plaque burden from the baseline to a 12 months coronary computed tomography angiography exam
Proportion of patients adherent to statin (%) | 12 months
  Assessed with questionnaire at 12 months follow-up
Change in high-sensitive CRP | 12 months
  Assessed by measurement of high-sensitive CRP level (mg/L) in blood samples at baseline and 12 months follow-up
Change in HbA1c | 12 months
  Assessed by measurement of HbA1c (mmol/mol) in blood samples at baseline and 12 months follow-up
Change in total-cholesterol levels | 12 months
  Assessed by measurement of total cholesterol levels (mmol/L) blood samples at baseline and 12 months follow-up
Proportion of patients in whom target LDL was reached (<1.8 mmol/L and ≤ 50% reduction relative to the non-treated LDL level) | 12 months
  Assessed with blood samples at baseline and 12 months follow-up, and preferably at 3 months
Change in dietary, exercise, and smoking habits | 12 months
  Assessed with questionnaire (based on national questionnaire every fourth year: "How are you?" (Hvordan har du det?)) at 12 months follow-up
Change in Angina and Quality of Life-scores | 12 months
  Assessed with questionnaire (based on HeartQoL and SAQ7) at baseline and12 months follow-up
Adverse clinical events (%) | 12 months
  Assessed by electronic patient records
Change in blood pressure | 12 months
  Unit of measure: mmHg. Assessed at 12 months follow-up
Change in Body Mass Index | 12 months
  Assessed at 12 months follow-up. Unit of measure kg/m2
Use of cardiovascular medication | 12 months
  Assessed by Electronic patient records and Shared Medication Record at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne L Nørgaard, Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Gødstrup Hospital, Gødstrup, Jutland
  - Aalborg University Hospital, Aalborg
  - Bjarne L Nørgaard, Aarhus
  - Hospital of South West Jutland, Esbjerg
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulasingam A, Laustsen S, Busk M, Sand NR, Winther S, Kragholm K, Hammid O, Pedersen KB, Vedsted P, Kanstrup H, Mortensen MB, Grove EL, Jensen JM, Norgaard BL. Rationale and design of VICAD-RISK study: Visualization of coronary artery disease for modification of risk factors. Am Heart J. 2025 Sep;287:16-23. doi: 10.1016/j.ahj.2025.04.002. Epub 2025 Apr 3. PMID 40187715